CLINICAL TRIAL: NCT04480034
Title: Laparoscopic Bariatric Surgery During Phase 2-3 Covid-19 Pandemic in Italy: a Multicenter, Prospective, Observational Study.
Brief Title: Obesity Surgery During 2020 Italian Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Ospedaliera di Padova (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); IRCCS Policlinico S. Donato (Other); University of Rome Tor Vergata (Other); A.O.U. Città della Salute e della Scienza (Other); Humanitas Clinical and Research Center (Other); Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, MD, PhD, Full Professor of Surgery, University of Roma La Sapienza
Other Study IDs: 008758/27.05.2020
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Bariatric Surgery Candidate; Covid19; Complication of Surgical Procedure; Pneumonia, Viral; Viral Infection; Obesity, Morbid; Safety Issues; Readmission
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Virus Diseases; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Group Pisa: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit UOC Chirurgia Bariatrica, Azienda Ospedaliera Universitaria Pisana, Pisa, Italy (Head Prof. Marco Anselmino) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Padova: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit UOSD Week Surgery, Azienda Ospedaliera, Università di Padova, Italy (Head Dr. Mirto Foletto) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Bologna: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit Chirurgia Bariatrica, Azienda Ospedaliera Universitaria di Bologna, Italy (Head Dr. Paolo Bernante) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Bergamo: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit UOC Chirurgia Generale e Oncologica, Policlinico San Marco di Zingonia, Bergamo, Italy (Head Prof. Stefano Olmi) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Tor Vergata: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit U.O.S.D. Chirurgia Mininvasiva e dell'Apparato Digerente, Università Tor Vergata, Rome, Italy (Head Prof. Paolo Gentileschi) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Torino: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit Dipartimento di Scienze Chirurgiche, Azienda Ospedaliera Universitaria Citta della Salute e della Scienza, Università di Torino, Italy (Head Prof. Mario Morino) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Milano: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit UO di Chirurgia Bariatrica, Humanitas Research Hospital, Rozzano, Milano, Italy (Head Dr. Giuseppe Marinari) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures
- Group Rome: All the bariatric cases (all laparoscopic bariatric procedures) performed during the period July/December 2020 in the unit UOC Chirurgia Generale & Bariatric Center of Excellence IFSO-EC, University La Sapienza of Rome, Italy (Head Prof. Gianfranco Silecchia) will be collected in a prospective database, to monitor the postoperative course.
  Interventions: Procedure: Bariatric procedures

INTERVENTIONS:
Procedure: Bariatric procedures — All standard, laparoscopic bariatric procedures endorsed by SICOB (Società Italiana della Chirurgia dell'Obesità, Italian Society of Obesity Surgery) and by IFSO (International Federation of the Societies of Obesity Surgery), will be considered: sleeve gastrectomy, R-en-Y gastric bypass, one anastomosis gastric bypass, single anastomosis duodeno-ileal bypass with sleeve. The selection criteria for the surgery candidates will comply to the latest guidelines for bariatric surgery endorsed by SICOB, IFSO and EAES (European Association of Endoscopic Surgery). All the participating centers will follow the usual recruitment protocol. Restart of the bariatric elective surgery is based on the guidelines of SICOB for the bariatric surgery restart in Italy during the COVID-19 phase 2-3 of endemics.

SUMMARY:
The first person-to-person Coronavirus disease (COVID-19) transmission in Italy was reported on Feb 21st, 2020, causing one of the most massive outbreak in Europe so far that stopped immediately all elective surgical procedures. Bariatric surgery represents the most effective treatment to obtain an important, long-term weight loss and comorbidities' resolution, including respiratory disorders. A sensitive decrease of epidemic has been observed lately and a gradual and progressive stop of the lockdown (phase 2-3) was planned, when the virus is supposed to be under control and protocols are guiding the restart of the elective bariatric surgery. Several questions are currently open: Laparoscopic bariatric surgery is safe in the phase 2-3? What's the expected complications rate? The actual hospital protocols are effective to minimize the risk of postoperative COVID-19 infection? Aim: to analyse results of bariatric surgery during phase 2-3 COVID-19 pandemic in Italy. Primary end point: 30 days COVID-19 infection, mortality and complications. Secondary end points: readmission rate 30 days, reoperations for any reason related to surgery. Study design: prospective multicenter observational. Setting: Italian National Health Service 8 high-volume bariatric centres. Enrollment criteria: No previous Covid-19 infection; Primary, standard IFSO approved bariatric procedures; No concomitant procedure; No previous major abdominal surgery; >18<60 years old; Compensated comorbidities; Official SICOB's surgical informed consent given, including COVID-19 addendum; Adherence to very restrictive protocols regarding: hospital admission, management of in-hospital patients and after discharge. Follow-up: scheduled outpatient visit 30th postoperative day. Data evaluation: all the cases performed during July/December 2020 will be collected in a prospective database. Patients operated during the period July/December 2019 in the same centers will be considered comparative group (control). Expected results: Transparent information to the patients, and the introduction of the COVID-19 protocol concerning patients and health-professionals protection, should guarantee a safe restart of bariatric surgery in Italy. The network of 8 high-volume centers sharing information and protocols in this "unexplored" period will be a guarantee for patients' safety. Bariatric surgery should induce a postoperative amelioration of the comorbidities reducing the risks in case of a second outbreak.

DETAILED DESCRIPTION:
Background Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) . The disease was first identified in December 2019 in Wuhan, the capital of China's Hubei province, and has since spread globally, resulting in the ongoing 2019-20 coronavirus pandemic . As of 08.05.2020, more than 3.91 million cases have been reported across 185 countries and territories, resulting in more than 218,000 deaths. More than 1.344.000 people have recovered . Even though there are very few available data on BMI for patients with COVID-19 infections, the role of obesity in the COVID-19 epidemic must not be ignored. A recent study on patients admitted in China for pneumonia from SARS-CoV-2, showed that obesity is associated with higher risks to develop severe pneumonia, especially in men . Obesity plays an important role in the pathogenesis of COVID-19 infection . In fact, the immune system, which is a key player in the pathogenesis of COVID-19, also plays an important role in obesity-induced adipose tissue inflammation. This inflammation of adipose tissue results in metabolic dysfunction potentially leading to dyslipidaemia, insulin resistance, type 2 diabetes mellitus, hypertension, and cardiovascular disease. A systematic review and meta-analysis demonstrated that severe obesity (body mass index BMI ≥ 40 kg/m2) represents a major risk factor of intensive care unit admission or death in individuals affected by H1N1 influenza . Thereafter, obesity is associated with a higher risk of infectious diseases, in particular of the respiratory tract.

There are a number of factors predisposing subjects with obesity to viral infections. These factors include low-grade chronic inflammation with hyper-production of pro-inflammatory cytokines, reduced natural killer (NK) cell number and activity, altered CD4:CD8T cell balance, impaired response to antigen stimulation and high expression of adipocyte angiotensin type 1 and 2 receptors.

Furthermore, obesity is associated with, and responsible for, comorbidity conditions that may represent risk factors for serious COVID-19 infection (i.e. type II diabetes, ischemic cardiac disease, etc.). Extra attention and precautions for patients with obesity during this epidemic is recommended. Whenever COVID-19 infection is suspected, screening must be systematic, particularly if the patient has obesity.

So far, bariatric surgery represents the most effective treatment to obtain a long-term meaningful weight reduction and resolution of comorbidities including respiratory disorders. In a very large case series study including 56277 subjects who underwent bariatric surgery in the United States, the overall risk of developing common infectious diseases including respiratory infections decreased significantly in men during the first two years after surgery (aOR, 0.69 [95% CI, 0.60-0.79]; P<0.001).

The first person-to-person transmission in Italy was reported on February 21st, 2020, in Lombardy region, the most crowded and rich region in Italy, causing the most massive Covid-19 outbreak in Europe so far. First positive cases of Sars-Co-v-2 were registered in Italy by 29th of January 2020. The COVID-19 outbreak stopped all elective surgical procedures by 9th of March, including bariatric/metabolic surgery except emergency conditions as suggested by recent IFSO recommendations . All elective surgical and endoscopic cases for metabolic and bariatric surgery should be postponed during the phase one outbreak. This would minimize risks to both patient and healthcare team, as well as reducing the utilization of unnecessary resources, such as beds, ventilators and personal protective equipment (PPE). In addition, postponing these services will minimize potential exposure of the COVID-19 virus to unsuspecting healthcare providers and patients.

To understand what could have been the impact of operating a population at risk of infection without specific precautions, we gathered a group of eight high-volume Italian bariatric centers, which performed 840 laparoscopic bariatric procedures during January and February 2020. Five are located in regions with high infection rates (Lombardy, Veneto, Piedmont, Emilia Romagna), and 3 are in areas with infection rate close to the Italian average (Tuscany, Lazio). A structured phone interview was administered to all patients operated during that period. We found five infections (5.9 cases out of 1000 inhabitants), four in Lombardy, and one in Veneto. The overall rate of infection on May 2, 2020, was similar in the 2 regions, 7.19 out of 1.000 inhabitants . Among infected patients, 2 had mild symptoms and home care, and three were hospitalized for fever and dyspnea; none died. Four out of five cases were over 60 years, all were female, and 3 out of 5 cases, reported an extra-hospital contact with positive COVID-19 people. All 5 cases healed eventually, with a negative swab.

During the last days of April 2020, a sensitive decrease of epidemic has been observed in Italy and Government planned a gradual and progressive stop of the lockdown (the so-called phase 2). That means the start of a new period when the virus is supposed to be under control and protocol are coming in the National Health Care System (SSN) to restart the elective surgical practice.

Several open questions are currently waiting the answers useful for the settlement of the management of obese patients, considering bariatric surgery effective for weight loss and co-morbidity control as well protective against eventual recurrent outbreak.

* Laparoscopic bariatric surgery is safe in the phase 2 outbreak?
* What's the expected complication rate of laparoscopic bariatric surgery in COVID-19 phase 2?
* The hospital protocols are effective to minimize the risk of postoperative Covid 19 infection after elective bariatric surgery in selected patients? Aim: to analyze results of laparoscopic bariatric surgery during phase 2 COVID-19 pandemic in Italy.

Primary end point: 30 days COVID-19 infection, mortality and complications. Secondary end points: readmission rate 30 days, reoperations for any reason related to bariatric surgery.

Study design: prospective multicenter observational Time interval: 12 months (July 2020 - May 2021): recruitment and therapy July 2020-December 2020, follow-up January 2021, data collection and analysis, manuscript preparation and publication Feb-May 2021).

Setting: Italian National Health Service' high-volume bariatric centres, academic hospitals.

Hospital admission protocol

1. Two to three days before admission, a doctor must interview the patient by telephone with the following questionnaire:

   * Did you have fever (threshold value > 37.5ºC / 99.5ºF), especially in the last 48 hours?
   * Do you have any new respiratory symptoms, especially when you walk?
   * Do you have other symptoms: vomiting, diarrhea, conjunctivitis, changes in smell, or taste, osteoarticular pain, excessive fatigue?
   * Have you had contact in the last two weeks with a confirmed case (clinical diagnosis - positive swab) of COVID-19?
2. 24-48 hours before hospitalization, the patient must arrive at the hospital: outside the hospital, the medical staff must repeat the interview as above and must swab the patient. In the case of a positive swab, surgery must be suspended. In the case of negativity, the patient must receive and sign a specific COVID-19 consent, and the operation can be carried out, with hospitalization on the same day of the procedure.

These procedures are in line with international and national guidelines for the screening of patients before entry the hospital (12) Screening at admission

1. Standard interview (National accepted Covid-19 questionnaire, see attachment 1)
2. Fever check
3. Chest X-ray / Thoracic CT scan Surgical informed consent

1. SICOB approved informed consent for standard bariatric procedures (2014 version); 2. A modified informed consent including the risk of COVID-1919 infection, will be adopted and added by all centers to the standard, above listed official consent: "I am aware that this bariatric procedure may lead to an increase in the possibility of contracting the COVID-19 infection, due to the general situation currently present, with a possible further increase in postoperative complications. I am also aware that, following the intervention, I will have to undergo a 14-day postoperative quarantine period, I will have to measure the temperature twice a day, I will be prohibited from traveling and traveling. The first postoperative check-up will be performed at the end of this period, unless complications related to surgery arise." Operating Room (OR) protocol

* For surgeon standard personal protective equipment (PPE) plus N95 mask
* For anesthesiologists and nurses who manage the airways and gastric bougie positioning, we recommend using N99 mask, face shield, single-use waterproof gown, and double gloves
* At the end of each procedure, every PPE must be changed
* Restrict access to people in OR
* Expert surgeons and anesthesiologists must perform the procedures to minimize the OR occupation time.
* A smoke evacuator system should be employed to avoid aerosol contamination; in the alternative, a filter must be connected to the exsufflation system.
* A negative pressure in the OR is not mandatory, but it is crucial to allow enough time between cases for complete room air exchange. In case the OR had been used for intensive care during phase 1 pandemic, proper sanitization is required.

Management of in-hospital patients

* No Covid-19 hospital/section should be used for elective bariatric surgery.
* Standard PPE for staff is mandatory.
* Social distance must be respected even in case of post-surgical mobilization; patients should always wear a surgical mask.
* Each patient should have a single room, or in the case of a large room, he must be assigned a suitable space to comply with the laws in force on social distancing.
* ERAS protocol is welcomed whenever is possible.

After discharge:

* In case of intra-hospital contact with Covid-19 patient or healthcare professional, 14 days self-quarantine after discharge is mandatory
* Home physical activity (same proposed program for all groups)
* Implement Oral supplementation (proposed recommendation for all groups)
* Low dose heparin for at least three weeks (proposed treatment for all groups)
* After 7 and 15 days the patients receive a follow-up phone with specific questions about Covid-19 (attached structured phone interview) Follow-up: Scheduled outpatient visit: 30 postoperative day.

ELIGIBILITY:
Inclusion Criteria:

1. Primary bariatric surgery;
2. Compensated DMT2;
3. Controlled hypertension;
4. Patients with OSAS can only be admitted if therapy with home CPAP is effective
5. Laparoscopic standard bariatric procedure;
6. Procedure duration less than 120 minutes;
7. Official SICOB's surgical informed consent given, including Covid-19 addendum.

Exclusion Criteria:

* previous Covid-19 infection;
* patients who may need an extended stay or intensive care (BMI > 60).
* concomitant procedure;
* previous major abdominal surgery

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Since July 2020, all the bariatric cases performed in the 8 participating centers will be collected in a prospective database, to monitor the postoperative course of the patients until WHO will declare the end of the pandemic, in order to determine the incidence of Sars-Cov-2 infection after bariatric surgery.
  All the data will be collected anonymously on a database by an independent data manager. The results will be evaluated in January 2021. As comparative group will be considered the patients operated during the period July/December 2019 in the same centers
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative COVID-19 infection | 30 postoperative days
  Postbariatric surgery COVID-19 infection, mortality and complications

SECONDARY OUTCOMES:
Complications related to bariatric surgery | 30 postoperative days
  Complications, reoperations for any reason related to bariatric surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University La Sapienza of Rome, Department of Medico-Surgical Sciences and Biotechnologies, Latina, LT, Italy

IPD SHARING:
Plan to Share IPD: Yes
All the data will be collected anonymously on a database by an independent data manager. All participants will have access to all recorded data through independent web access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: restricted access, based on username and password dedicated for every group
URL: https://test-chirurgiabariatricadurantecovid.pantheonsite.io/

REFERENCES:
- [Result] Hui DS, I Azhar E, Madani TA, Ntoumi F, Kock R, Dar O, Ippolito G, Mchugh TD, Memish ZA, Drosten C, Zumla A, Petersen E. The continuing 2019-nCoV epidemic threat of novel coronaviruses to global health - The latest 2019 novel coronavirus outbreak in Wuhan, China. Int J Infect Dis. 2020 Feb;91:264-266. doi: 10.1016/j.ijid.2020.01.009. Epub 2020 Jan 14. No abstract available. PMID 31953166
- [Result] Chen Q, Zheng Z, Zhang C, Zhang X, Wu H, Wang J, Wang S, Zheng C. Clinical characteristics of 145 patients with corona virus disease 2019 (COVID-19) in Taizhou, Zhejiang, China. Infection. 2020 Aug;48(4):543-551. doi: 10.1007/s15010-020-01432-5. Epub 2020 Apr 28. PMID 32342479
- [Result] Kassir R. Risk of COVID-19 for patients with obesity. Obes Rev. 2020 Jun;21(6):e13034. doi: 10.1111/obr.13034. Epub 2020 Apr 13. No abstract available. PMID 32281287
- [Result] Honce R, Schultz-Cherry S. Impact of Obesity on Influenza A Virus Pathogenesis, Immune Response, and Evolution. Front Immunol. 2019 May 10;10:1071. doi: 10.3389/fimmu.2019.01071. eCollection 2019. PMID 31134099
- [Result] Kornum JB, Norgaard M, Dethlefsen C, Due KM, Thomsen RW, Tjonneland A, Sorensen HT, Overvad K. Obesity and risk of subsequent hospitalisation with pneumonia. Eur Respir J. 2010 Dec;36(6):1330-6. doi: 10.1183/09031936.00184209. Epub 2010 Mar 29. PMID 20351023
- [Result] Shapouri-Moghaddam A, Mohammadian S, Vazini H, Taghadosi M, Esmaeili SA, Mardani F, Seifi B, Mohammadi A, Afshari JT, Sahebkar A. Macrophage plasticity, polarization, and function in health and disease. J Cell Physiol. 2018 Sep;233(9):6425-6440. doi: 10.1002/jcp.26429. Epub 2018 Mar 1. PMID 29319160
- [Result] Cheng CI, Chen PH, Lin YC, Kao YH. High glucose activates Raw264.7 macrophages through RhoA kinase-mediated signaling pathway. Cell Signal. 2015 Feb;27(2):283-92. doi: 10.1016/j.cellsig.2014.11.012. Epub 2014 Nov 14. PMID 25446262
- [Result] Torres-Castro I, Arroyo-Camarena UD, Martinez-Reyes CP, Gomez-Arauz AY, Duenas-Andrade Y, Hernandez-Ruiz J, Bejar YL, Zaga-Clavellina V, Morales-Montor J, Terrazas LI, Kzhyshkowska J, Escobedo G. Human monocytes and macrophages undergo M1-type inflammatory polarization in response to high levels of glucose. Immunol Lett. 2016 Aug;176:81-9. doi: 10.1016/j.imlet.2016.06.001. Epub 2016 Jun 4. PMID 27269375
- [Result] Sun JC, Beilke JN, Lanier LL. Adaptive immune features of natural killer cells. Nature. 2009 Jan 29;457(7229):557-61. doi: 10.1038/nature07665. Epub 2009 Jan 11. PMID 19136945
- [Result] van der Weerd K, Dik WA, Schrijver B, Schweitzer DH, Langerak AW, Drexhage HA, Kiewiet RM, van Aken MO, van Huisstede A, van Dongen JJ, van der Lelij AJ, Staal FJ, van Hagen PM. Morbidly obese human subjects have increased peripheral blood CD4+ T cells with skewing toward a Treg- and Th2-dominated phenotype. Diabetes. 2012 Feb;61(2):401-8. doi: 10.2337/db11-1065. Epub 2012 Jan 6. PMID 22228716
- [Result] Smith AG, Sheridan PA, Harp JB, Beck MA. Diet-induced obese mice have increased mortality and altered immune responses when infected with influenza virus. J Nutr. 2007 May;137(5):1236-43. doi: 10.1093/jn/137.5.1236. PMID 17449587
- [Result] Mauro C, Smith J, Cucchi D, Coe D, Fu H, Bonacina F, Baragetti A, Cermenati G, Caruso D, Mitro N, Catapano AL, Ammirati E, Longhi MP, Okkenhaug K, Norata GD, Marelli-Berg FM. Obesity-Induced Metabolic Stress Leads to Biased Effector Memory CD4+ T Cell Differentiation via PI3K p110delta-Akt-Mediated Signals. Cell Metab. 2017 Mar 7;25(3):593-609. doi: 10.1016/j.cmet.2017.01.008. Epub 2017 Feb 9. PMID 28190771
- [Result] Walls AC, Park YJ, Tortorici MA, Wall A, McGuire AT, Veesler D. Structure, Function, and Antigenicity of the SARS-CoV-2 Spike Glycoprotein. Cell. 2020 Apr 16;181(2):281-292.e6. doi: 10.1016/j.cell.2020.02.058. Epub 2020 Mar 9. PMID 32155444
- [Result] Schling P, Mallow H, Trindl A, Loffler G. Evidence for a local renin angiotensin system in primary cultured human preadipocytes. Int J Obes Relat Metab Disord. 1999 Apr;23(4):336-41. doi: 10.1038/sj.ijo.0800821. PMID 10340809
- [Result] Engeli S, Negrel R, Sharma AM. Physiology and pathophysiology of the adipose tissue renin-angiotensin system. Hypertension. 2000 Jun;35(6):1270-7. doi: 10.1161/01.hyp.35.6.1270. PMID 10856276
- [Result] Onder G, Rezza G, Brusaferro S. Case-Fatality Rate and Characteristics of Patients Dying in Relation to COVID-19 in Italy. JAMA. 2020 May 12;323(18):1775-1776. doi: 10.1001/jama.2020.4683. No abstract available. PMID 32203977
- [Result] Bornstein SR, Dalan R, Hopkins D, Mingrone G, Boehm BO. Endocrine and metabolic link to coronavirus infection. Nat Rev Endocrinol. 2020 Jun;16(6):297-298. doi: 10.1038/s41574-020-0353-9. PMID 32242089
- [Result] Maggard MA, Shugarman LR, Suttorp M, Maglione M, Sugerman HJ, Livingston EH, Nguyen NT, Li Z, Mojica WA, Hilton L, Rhodes S, Morton SC, Shekelle PG. Meta-analysis: surgical treatment of obesity. Ann Intern Med. 2005 Apr 5;142(7):547-59. doi: 10.7326/0003-4819-142-7-200504050-00013. PMID 15809466
- [Result] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Nanni G, Castagneto M, Bornstein S, Rubino F. Bariatric-metabolic surgery versus conventional medical treatment in obese patients with type 2 diabetes: 5 year follow-up of an open-label, single-centre, randomised controlled trial. Lancet. 2015 Sep 5;386(9997):964-73. doi: 10.1016/S0140-6736(15)00075-6. PMID 26369473
- [Result] Capoccia D, Guida A, Coccia F, Guarisco G, Testa M, Leonetti F, Silecchia G. Weight Regain and Diabetes Evolution After Sleeve Gastrectomy: a Cohort Study with over 5 Years of Follow-Up. Obes Surg. 2020 Mar;30(3):1046-1051. doi: 10.1007/s11695-019-04350-0. PMID 31853861
- [Result] Sjostrom L. Review of the key results from the Swedish Obese Subjects (SOS) trial - a prospective controlled intervention study of bariatric surgery. J Intern Med. 2013 Mar;273(3):219-34. doi: 10.1111/joim.12012. Epub 2013 Feb 8. PMID 23163728
- [Result] Goto T, Hirayama A, Faridi MK, Camargo CA Jr, Hasegawa K. Association of Bariatric Surgery With Risk of Infectious Diseases: A Self-Controlled Case Series Analysis. Clin Infect Dis. 2017 Oct 15;65(8):1349-1355. doi: 10.1093/cid/cix541. PMID 28637274
- [Result] Sharma P, McCarty TR, Ngu JN, O'Donnell M, Njei B. Impact of bariatric surgery in patients with HIV infection: a nationwide inpatient sample analysis, 2004-2014. AIDS. 2018 Sep 10;32(14):1959-1965. doi: 10.1097/QAD.0000000000001915. PMID 30157083
- [Result] Yang W, Wang C, Shikora S, Kow L. Recommendations for Metabolic and Bariatric Surgery During the COVID-19 Pandemic from IFSO. Obes Surg. 2020 Jun;30(6):2071-2073. doi: 10.1007/s11695-020-04578-1. No abstract available. PMID 32291701
- [Result] Di Lorenzo N, Antoniou SA, Batterham RL, Busetto L, Godoroja D, Iossa A, Carrano FM, Agresta F, Alarcon I, Azran C, Bouvy N, Balague Ponz C, Buza M, Copaescu C, De Luca M, Dicker D, Di Vincenzo A, Felsenreich DM, Francis NK, Fried M, Gonzalo Prats B, Goitein D, Halford JCG, Herlesova J, Kalogridaki M, Ket H, Morales-Conde S, Piatto G, Prager G, Pruijssers S, Pucci A, Rayman S, Romano E, Sanchez-Cordero S, Vilallonga R, Silecchia G. Clinical practice guidelines of the European Association for Endoscopic Surgery (EAES) on bariatric surgery: update 2020 endorsed by IFSO-EC, EASO and ESPCOP. Surg Endosc. 2020 Jun;34(6):2332-2358. doi: 10.1007/s00464-020-07555-y. Epub 2020 Apr 23. PMID 32328827